CLINICAL TRIAL: NCT03690817
Title: The Link Between Hearing Loss, Vestibular Loss and Cognitive Performance: Cross-sectional Data in Patients With Bilateral Vestibulopathy
Brief Title: Hearing Loss, Vestibular Loss and Cognitive Performance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Ethisch Comité, UZA, Principal Investigator, University Hospital, Antwerp
Other Study IDs: 16/42/426
Record Dates: First submitted 2018-08-27; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Vestibular Disorder
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bilateral vestibulopathy: Patients with bilateral vestibulopathy, according to the Barany Criteria (2017, Strupp).
  Interventions: Behavioral: RBANS-H, virtual Morris Water Maze
- Healthy controls: Subjects without vestibular or neurological diseases (DHI<5), and with normal hearing thresholds according to their age.
  Interventions: Behavioral: RBANS-H, virtual Morris Water Maze

INTERVENTIONS:
Behavioral: RBANS-H, virtual Morris Water Maze — Cognitive tasks for respectively: general cognition and spatial cognition

SUMMARY:
Hearing loss is an established independent risk factor for dementia. Likewise, recent research demonstrated cognitive deficits in subjects with vestibular loss. However, in these studies data have not been adjusted for the hearing status of the enrolled study subjects. As hearing loss prevalence is high in patients with vestibular loss, this could be a major confounder. Therefore, in this study the investigators investigate cognition in patients with bilateral vestibulopathy with and without hearing loss. The investigators adjust data for the hearing status of the patients to explore the link between hearing loss, vestibular loss and cognition.

ELIGIBILITY:
Inclusion criteria for BVP patients were:

1. Bilaterally reduced vestibular function, as defined by the Bárány Criteria for BVP (Michael Strupp 2017):

   * horizontal angular VOR gain < 0.6 measured by the vHIT, and/or
   * reduced caloric response (sum of bithermal, 30° and 44°, max. peak slow phase velocity (SPV) on each side < 6°/sec), and/or
   * reduced horizontal angular VOR gain < 0.1 upon sinusoidal stimulation on a rotatory chair. At our clinic rotatory chair tests are performed using sinusoidal rotation (0.05 Hertz) with a peak velocity of 60°/sec (Van der Stappen A 2000).
2. Disease duration of BVP > 6 months.

Healthy controls (HC). Only subjects with no history of vertigo, scores <5 on the Dizziness Handicap Inventory (DHI) and normal hearing thresholds at 0.25 - 8 kHz, based on age and sex (defined by the BS 6951:1988, EN 27029:1991 and ISO 7029-1984 standards), were enrolled in the study.

For both BVP patients and HC the following additional inclusion criteria were applied: 1) Age ≥ 18 years; 2) Fluency in Dutch; 3) No history of neurological diseases (e.g. dementia, Parkinson's disease, cerebrovascular accident, etc.); 4) Absence of clinical signs indicating dementia or mild cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with bilateral vestibulopathy, which was confirmed by vestibular testing, were enrolled in the patient group. Healthy controls with normal hearing and vestibular system were used to compare cognitive outcome measures with. Correction were made for age, sex, education and computer usage.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
The Repeatable Battery for the Assessment of Neuropsychological Status for Hearing Impaired Individuals (RBANS-H): total score | 2 years
  General cognitive assessment, cfr. Claes et al 2016. The total-score is standardized with a mean of 100 and a standard deviation of 15. The higher the total score, the better the cognition of the participant.
Virtual Morris Water Maze performance | 2 years
  Spatial cognition assessment, cfr. Hamilton. Path length and latency are recorded, the higher the worse the spatial cognition of the participant.

SECONDARY OUTCOMES:
The Repeatable Battery for the Assessment of Neuropsychological Status for Hearing Impaired Individuals (RBANS-H): index scores | 2 years
  Cfr. Claes et al 2016. The subscale are standardized with a mean of 100 and standard deviation of 15. The higher the score, the better the performance on a specific subdomain of cognition (attention, immediate memory, delayed memory, visuospatial and language)

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peetermans O, Dobbels B, Mertens G, Moyaert J, van de Berg R, Vanderveken O, Van de Heyning P, Perez Fornos A, Guinand N, Lammers MJW, Van Rompaey V. Sound localization in patients with bilateral vestibulopathy. Eur Arch Otorhinolaryngol. 2022 Dec;279(12):5601-5613. doi: 10.1007/s00405-022-07414-7. Epub 2022 May 10. PMID 35536383